CLINICAL TRIAL: NCT00928044
Title: The Impact of Gynecological Surgery on Ovarian Function in Women of Reproductive Age: Postoperative Changes of Serum Anti-Müllerian Hormone
Brief Title: The Impact of Gynecological Surgery on Ovarian Function in Women of Reproductive Age: Postoperative Changes of Serum Anti-Müllerian Hormone (AMH)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: DooSeok Choi, Samsung Medical Center
Other Study IDs: 2008-01-050
Record Dates: First submitted 2009-06-24; First posted 2009-06-25 (Estimated); Last update posted 2009-06-25 (Estimated); Status verified 2009-06

CONDITIONS: Gynecologic Operations; Anti-Mullerian Hormone; Ovarian Reserve

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample was taken before and in 1 week, 1 month and 3 months after surgery for operation group or at the time of screening for control group, and transvaginal ultrasonography was performed with AMH sampling.
  After collection of blood, serum was stored at -70ºC until the measurement of AMH level. Serum levels of AMH were determined by an enzyme-linked immunosorbent assay using commercial kit (Beckman Coulter Inc., Paris, France)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- control groups: They had regular menstrual cycles and no history of pelvic surgery. None had any endocrine disorders (e.g. PCOS) and received any kind of medication that could affect the results within the preceding 6 months, and any woman who had a suspected pathologic lesion in the ovary or menopausal symptoms was excluded.
- operation group: 1. They had regular menstrual cycles and no history of pelvic surgery. None had any endocrine disorders (e.g. PCOS) and received any kind of medication that could affect the results within the preceding 6 months, and any woman who had a suspected pathologic lesion in the ovary or menopausal symptoms was excluded. 2. Operations were performed for benign ovarian tumors, leiomyoma or adenomyosis

SUMMARY:
Besides the removal of lesions, the purpose of surgeries has been extended to the improvement of quality of life after procedures. Minimally invasive surgeries enabled women to experience less pain, less hospital days. It is important to maintain the ovarian function because ovarian hormones have protective effects about bone and cardiovascular diseases. Until now many operation techniques for preserving ovarian function were used in gynecological field, however, how much these methods affect on ovarian function is seldom known. For the evaluation of remained ovarian function, ultrasound examination is useful method. However, it might take several months till one can determine ovarian function and could not exactly evaluate ovarian reserve. Until now, there have been controversies regarding ovarian function after gynecological surgeries. These inconsistent results might derive from the methods for assessing ovarian function because serum gonadotropins and sex steroids levels vary according to the menstrual cycle.

In this aspect, anti-Müllerian hormone (AMH) has recently been advocated as a good marker for ovarian reserve. AMH is one of the TGF-beta superfamily and induces the regression of Müllerian duct. Studies with AMH showed no significant variation throughout the menstrual cycle and cycle-to-cycle consistency, therefore, it will provide more reliable data on the changes of ovarian reserve after operations.

DETAILED DESCRIPTION:
Premenopausal women were enrolled and were allocated into two groups; operation and control group. Operations were performed for benign ovarian tumors, leiomyoma or adenomyosis. All eligible women were identified from the Samsung Medical Center. Written informed consent was obtained from all subjects and the study was approved by the Institutional Review Board of Samsung Medical Center.

A complete medical history was taken, and physical and gynecological examinations were performed at baseline. Data included information on age, menstrual cycle, parity, weight, height, and BMI. The follow-up length was 3 months. Blood sample was taken before and in 1 week, 1 month and 3 months after surgery for operation group or at the time of screening for control group, and transvaginal ultrasonography was performed with AMH sampling.

After collection of blood, serum was stored at -70ºC until the measurement of AMH level. Serum levels of AMH were determined by an enzyme-linked immunosorbent assay using commercial kit (Beckman Coulter Inc., Paris, France). The detection limit of the assay was 0.14 ng/mL, and the intra- and inter-assay coefficients of variation were 12.3% and 14.2%, respectively.

Ultrasonographic examination was performed using the ALOKA prosound SSD-3500 (ALOKA, Wallingford, CT, USA) with a 7.5-MHz vaginal probe for color Doppler ultrasonography to assess the ovarian artery flow at the ovarian hilum. The pulsatile index (PI) and resistance index (RI) values were calculated according to the formula PI=[S-D]/mean and RI=[S-D]/S, where S was the peak systolic flow velocity; D was diastolic velocity; and the mean was the mean flow velocity. All examinations were conducted by the same investigator to minimize interobserver bias, and parameters were measured at least 3 times and the mean value was recorded.

Operations were performed by gynecologists in our center using the technique of laparoscopy-assisted vaginal or trans-abdominal approaches for hysterectomy and using oophorectomy or cystectomy method for ovarian disease.

Statistical analyses were performed using Statistical Analysis System (SAS Institute Inc., version 9.1, Enterprise Guide 3.0, Cary, NC, USA) and R (version 2.7.2) by a statistician in our hospital. The Fisher's exact test was used for frequency data. The variables presenting normal distribution were compared by t test or analysis of variance. For the variables which did not show normal distribution, the Kruskal-Wallis test or Wilcoxon test were used. A P-value <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* For both operation and control groups, women were eligible for inclusion if they had regular menstrual cycles and no history of pelvic surgery.

Exclusion Criteria:

* No endocrine disorders (e.g. PCOS).
* Received any kind of medication that could affect the results within the preceding 6 months.
* Any woman who had a suspected pathologic lesion in the ovary or menopausal symptoms.

Ages: 20 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Premenopausal women were enrolled and were allocated into two groups; operation and control group. Operations were performed for benign ovarian tumors, leiomyoma or adenomyosis. All eligible women were identified from the Samsung Medical Center. Written informed consent was obtained from all subjects and the study was approved by the Institutional Review Board of Samsung Medical Center.
  A complete medical history was taken, and physical and gynecological examinations were performed at baseline. Data included information on age, menstrual cycle, parity, weight, height, and BMI. The follow-up length was 3 months. Blood sample was taken before and in 1 week, 1 month and 3 months after surgery for operation group or at the time of screening for control group, and transvaginal ultrasonography was performed with AMH sampling.
Sampling Method: Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-01 (Estimated); Study Completion 2009-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: DooSeok Choi, MD, PhD, Principal Investigator — Samsung Medical Center